CLINICAL TRIAL: NCT04244929
Title: Clinical Evaluation of the Total Knee Prosthesis Persona Medial Congruent® With Preservation or Sacrifice of the Posterior Cruciate Ligament: a Multicentric Perspective Study
Brief Title: Multicenter Perspective Study: Clinical Evaluation of the Persona MC® With Preservation or Sacrifice of the PCL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: Persona-MC
Record Dates: First submitted 2020-01-20; First posted 2020-01-28 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Prosthesis Survival
MeSH Terms: conditions — Prosthesis Failure | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Intervention Model Description: Prospective, two arms, multicenter study that aims to involve up to 10 hospitals in Italy
Who Masked: Outcomes Assessor
Masking Description: The Co-Investigator who assesses the outcomes will be blind to the treatment group's allocation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PCL removal (Experimental): Patients will undergo surgery by sacrificing the PCL
  Interventions: Procedure: Total knee arthroplasty; Device: Persona Medial Congruent Knee Prosthesis implantation with Posterior Cruciate Ligament sacrifice
- PCL preservation (Active Comparator): Patients will undergo surgery with retaining the PCL
  Interventions: Procedure: Total knee arthroplasty; Device: Persona Medial Congruent Knee Prosthesis implantation with Posterior Cruciate Ligament retaining

INTERVENTIONS:
Procedure: Total knee arthroplasty — Total knee arthroplasty using standard anterior approach.
Device: Persona Medial Congruent Knee Prosthesis implantation with Posterior Cruciate Ligament retaining — Patients will be implanted with this medial pivoting knee prosthesis. Posterior Cruciate Ligament will be retained
  Arms: PCL preservation
Device: Persona Medial Congruent Knee Prosthesis implantation with Posterior Cruciate Ligament sacrifice — Patients will be implanted with this medial pivoting knee prosthesis. Posterior Cruciate Ligament will be sacrificed
  Arms: PCL removal

SUMMARY:
Prospective, multicenter study on the Total Knee Prosthesis available on the market "Persona Medial Congruent® knee".

Primary endpoint

-Evaluation of the survival of the implant after 5 years of follow-up

Secondary endpoints

* Evaluation of the survival of the implant at 10 years of follow up.
* Evaluation of clinical and radiographic outcomes in Italian patients undergoing total knee replacement with the Persona Medial Congruent® implant with sacrifice or retention of the posterior cruciate ligament (PCL)

DETAILED DESCRIPTION:
Prospective, multicenter study on the Total Knee Prosthesis available on the market "Persona Medial Congruent® knee" Up to 10 Italian centers will provide a maximum of 200 patients undergoing total knee replacement with Persona prosthesis and Medial Congruent® insert.

20 cases per center will be performed, 10 with posterior cruciate ligament sacrifice, 10 with posterior cruciate ligament preservation.

Patients will be recruited and enrolled in the study according to the inclusion and exclusion criteria specified below. In order to minimize the selection bias, patients will be enrolled consecutively; the first 10 patients will constitute a treatment group and the remaining 10 the complementary group.

Each patient will sign an informed consent for participation in the prospective study. The patients will be recruited at the Orthopedic and Traumatological Clinic 2nd of the Rizzoli Orthopedic Institute on an outpatient or hospitalization basis.

After the surgical treatment, the patient will continue his hospitalization at the Orthopedic and Traumatological Clinic 2nd of the Rizzoli Orthopedic Institute and, if deemed appropriate by the medical team, he will be discharged by planning the subsequent post-operative checks and diagnostic evaluations.

The data will be collected by investigators and provided to the Promoter center.

The Co-investigator who will evaluate the results will be blind to the assignment to the treatment group of the subjects in the study. The promoter of the study is the owner of the data and therefore responsible for data management. Study participants are identified with an identification code. All sensitive personal data will be stored in accordance with the current data privacy guidelines. All information will be treated with strict compliance with professional confidentiality standards. Participants will receive oral and written information relating to the processing of sensitive personal data.

The study is designed to have an alpha error of no more than 0.05. Based on an assumed 95% five-year survival, a sample size of n = 89 was calculated using SAS 9.4, Proc Power.

Assuming a 20% follow-up loss rate over five years, the study will enroll 100 patients in each patient group, then a total of 200 patients. The data collected from 200 patients (100 in each subgroup) will be archived in a descriptive way and will be the basis of all published study reports.

The categorical data (for example, gender) will be summarized using counts, percentages and the 95% confidence interval (CI), in the periods of interest. Continuous data, such as age, will be summarized using means, medians, standard deviation, minimum, maximum and 95% CI in the periods of interest. Implant survival and return to function will be summarized using the Kaplan-Meier method and presented as percentages and confidence intervals.

The expected duration of the study is 11 years, which corresponds to the time dedicated to the approval of the Ethics Committee, the enrollment of all patients, the completion of the 10-year follow-up, data analysis and preparation of the final report. The first 12 months will focus on patient enrollment. The study subjects will be involved from the moment of the intervention until the end of the 10-year follow-up (as per the current protocol 10 years FU ± 2 months).

ELIGIBILITY:
Inclusion Criteria:

* Patient qualifies for a primary total knee arthroplasty based on physical exam and medical history, including diagnosis of severe knee pain and disability due to at least one of the following:

  1. Rheumatoid arthritis, osteoarthritis, traumatic arthritis, polyarthritis
  2. Collagen disorders and/or avascular necrosis of the femoral condyle
  3. Post-traumatic loss of joint configuration, particularly when there is patellofemoral erosion, dysfunction or prior patellectomy
  4. Moderate valgus, varus, or flexion deformities
  5. The salvage of previously failed surgical attempts that did not include partial or total knee arthroplasty of the ipsilateral knee
* Patient is willing and able to complete scheduled study procedures and follow-up evaluations
* Independent of study participation, patient is a candidate for commercially available Persona MC knee implants. Patient is willing and able to complete scheduled follow-up evaluations as described in the Informed Consent.
* Patient has participated in the Informed Consent process and has signed the Ethics Committee approved 'Informed Consent'.

Exclusion Criteria:

* Patient is currently participating in any other surgical intervention studies or pain management studies
* Patient is unwilling or unable to give consent or to comply with the follow-up program.
* Patient meets exclusion criteria of the Instruction for Use Patients who have any condition which would in the judgement of the Investigator place the patient at undue risk or interfere with the study. Any patient who is institutionalized, or is a known drug abuser, a known alcoholic or anyone who cannot understand what is required of them.
* Previous history of infection in the affected joint and/or other local/systemic infection that may affect the prosthetic joint
* Insufficient bone stock on femoral or tibial surfaces
* Skeletal immaturity
* Neuropathic arthropathy
* Osteoporosis or any loss of musculature or neuromuscular disease that compromises the affected limb
* Stable, painless arthrodesis in a satisfactory functional position
* Severe instability secondary to the absence of collateral ligament integrity
* Rheumatoid arthritis accompanied by an ulcer of the skin or a history of recurrent breakdown of the skin
* Patient has a known or suspected sensitivity or allergy to one or more of the implant materials

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety based on implant survivorship at 5 years follow up | 72 months
  Implant survival will be evaluated by radiographic parameters on standard and long leg standing radiographs that indicate prosthesis mobilization (radiolucency lines, fracture, osteolysis)

SECONDARY OUTCOMES:
Evaluate the safety based on implant survivorship at 10 years follow up | 132 months
  Implant survival will be evaluated by radiographic parameters on standard and long leg standing radiographs that indicate prosthesis mobilization (radiolucency lines, fracture, osteolysis)
Evaluation of pain | 132 months
  Clinical evaluation addresses the state of the studied knee before and after the surgery with respect to pain (VAS scale).
Evaluation of medication taken by the patient | 132 months
  Clinical evaluation addresses the state of the studied knee before and after the surgery with respect to medications.
Evaluation of muscle strength | 132 months
  Clinical evaluation addresses the state of the studied knee before and after the surgery with respect to muscle strength, evaluated with a subjective scale by the investigator
Return to work | 132 months
  Additional information regarding the returning of the patient to work is collected at 3 or 6 months follow up
Patient Satisfaction Questionnaire | 132 months
  It is a patient-reported short questionnaire for evaluating patient satisfaction with the knee replacement surgery
Euro Quality of Life-5 Dimensions-5 Levels Health Questionnaire | 132 months
  It is completed by the patient and assesses his/her general health status. The EQ-5D is used to derive a quality of life index used for health economics considerations
Oxford Knee Score | 132 months
  It is a patient-reported form and consists of 12 questions on the influence of the knee (surgical side) on daily activities or pain.
American Knee Society Score | 132 months
  It is used to assess knee functionality by investigator. It consists of both a clinical and a functional score
Forgotten Joint Score | 132 months
  is completed by the patient and assesses his/her ability to forget about his/ her knee joint prior and after treatment
Adverse Event Report | 132 months
  is completed as needed for each complication which is noted. Each complication shall be examined again at the next follow-up visit and further documented on a separate form for each visit.
Explanted Device Form | 132 months
  collects information on revision surgeries for study subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Maria Marcheggiani Muccioli, MD, PhD, Principal Investigator — IRCCS Istituto Ortopedico Rizzoli
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sabatini L, Risitano S, Parisi G, Tosto F, Indelli PF, Atzori F, Masse A. Medial Pivot in Total Knee Arthroplasty: Literature Review and Our First Experience. Clin Med Insights Arthritis Musculoskelet Disord. 2018 Jan 4;11:1179544117751431. doi: 10.1177/1179544117751431. eCollection 2018. PMID 29326531
- [Background] Van Overschelde PP, Fitch DA. Patient satisfaction at 2 months following total knee replacement using a second generation medial-pivot system: follow-up of 250 consecutive cases. Ann Transl Med. 2016 Sep;4(18):339. doi: 10.21037/atm.2016.08.41. PMID 27761443
- [Result] Bourne RB, Chesworth BM, Davis AM, Mahomed NN, Charron KD. Patient satisfaction after total knee arthroplasty: who is satisfied and who is not? Clin Orthop Relat Res. 2010 Jan;468(1):57-63. doi: 10.1007/s11999-009-1119-9. PMID 19844772
- [Result] Nam D, Nunley RM, Barrack RL. Patient dissatisfaction following total knee replacement: a growing concern? Bone Joint J. 2014 Nov;96-B(11 Supple A):96-100. doi: 10.1302/0301-620X.96B11.34152. PMID 25381418